CLINICAL TRIAL: NCT02454010
Title: A Phase 1 Dose-escalation Study of Radio- Labeled Antibody, FF-21101(90Y) for the Treatment of Advanced Cancer
Brief Title: A Dose Escalation Study of Radio-labeled Antibody for the Treatment of Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujifilm Pharmaceuticals U.S.A., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FF21101US101
Record Dates: First submitted 2015-05-04; First posted 2015-05-27 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Lowest dose of FF-21101(90Y) (Experimental): In the therapeutic phase subjects in this cohort will receive one dose of radiolabeled FF21101
  Interventions: Biological: FF21101
- 2X Lowest dose of FF-21101(90Y) (Experimental): In the therapeutic phase subjects in this cohort will receive one dose of radiolabeled FF21101 that is 2X the lowest dose
  Interventions: Biological: FF21101
- 3X Lowest dose of FF-21101(90Y) (Experimental): In the therapeutic phase subjects in this cohort will receive one dose of radiolabeled FF21101 that is 3X the lowest dose
  Interventions: Biological: FF21101
- 4X Lowest dose of FF-21101(90Y) (Experimental): In the therapeutic phase subjects in this cohort will receive one dose of radiolabeled FF21101 that is 4X the lowest dose
  Interventions: Biological: FF21101
- 5X Lowest dose of FF-21101(90Y) (Experimental): In the therapeutic phase subjects in this cohort will receive one dose of radiolabeled FF21101 that is 5X the lowest dose
  Interventions: Biological: FF21101
- Expansion Phase (Cohort 6), Ovarian (Experimental): In the expansion phase, subjects in this cohort will be diagnosed with epithelial ovarian, peritoneal or fallopian tube carcinoma and will receive a dose of 25 mCi/m2 FF-21101(90Y)
  Interventions: Biological: FF21101
- Expansion Phase (Cohort 7), Adv Tumors (Experimental): In the expansion phase, subjects in this cohort will be diagnosed with triple negative breast cancer (TNBC), head and neck squamous cell carcinoma (HNSCC), biliary cancer (cholangiocarcinoma or gall bladder carcinoma), pancreatic carcinoma, colorectal cancer and will receive a dose of 25 mCi/m2 FF-21101(90Y)
  Interventions: Biological: FF21101

INTERVENTIONS:
Biological: FF21101 — (90Y) radio-labeled FF21101 (therapeutic monoclonal antibody to P-cadherin expressed by the CDH3 gene)

SUMMARY:
The purpose of this study is to determine the safety and tolerability in subjects who receive FF-21101(111In) for dosimetry and FF-21101(90Y) for treatment of advanced solid tumors.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and tolerability in subjects who receive FF-21101(111In) for dosimetry and FF-21101(90Y) for treatment of advanced solid tumors. This is an open label study that will recruit approx 70 patients

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Histologically or cytologically confirmed advanced solid tumor malignancy, refractory or relapsed from prior therapy, or for whom no alternative therapy is available
* At least 4 weeks beyond the last chemotherapy (or ≥ 5 half-lives for targeted agents, whichever is shorter), radiotherapy, major surgery or experimental treatment and recovered from all acute toxicities (≤ Grade 1)
* Archival tumor sample available, or be willing to undergo a fresh tumor biopsy, prior to study
* At least one measurable disease site that meets target lesion requirements
* Adequate performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Life expectancy of ≥ 3 months
* Adequate hematologic parameters without ongoing transfusional support:
* Negative serum pregnancy test
* Ability to provide written informed consent

Exclusion Criteria:

* Previous radioimmunotherapy. Previous antibody-based therapy is allowed as long as ≥ 28 days has elapsed from last dose to study treatment.
* Prior radiation to > 30% of the red marrow or to maximal tolerable level for any organ
* Serious cardiac condition within the last 6 months
* Concomitant medication(s) that may cause QTc prolongation or induce Torsades de Pointes, with the exception of antimicrobials that are considered to be essential for care of the patient
* History of retinal degenerative disease, history of uveitis, history of retinal vein occlusion (RVO), or any eye condition that would be considered a risk factor for RVO or has medically relevant abnormalities identified on screening ophthalmologic examination
* Active central nervous system (CNS) malignant disease in subjects with a history of CNS malignancy. Subjects with stable, prior, or currently treated brain metastases are allowed.
* Known positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV)
* Known autoimmune disease
* Active infection requiring intravenous (IV) antibiotic usage within the last week prior to the dosimetry portion of the study
* Corticosteroid use within 2 weeks of study treatment
* Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence with study requirements or confound the interpretation of study results
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of radio-labeled FF21101 | 28 days
  measured by number of patients with adverse events leading to discontinuation or number of patients with dose limiting toxicity

SECONDARY OUTCOMES:
Number of patients achieving overall response using Response Evaluation Criteria in Solid Tumors (RECIST v. 1.1) | 8 weeks
  Overall response rates are defined as the number of patients achieving a best response of complete response [CR], partial response [PR], stable disease [SD], or progressive disease [PD])

OTHER OUTCOMES:
Number of patients expressing CDH3 (human cadherin 3/P-cadherin) as a predictor of clinical activity | Single sample taken at enrollment
  measurement of CDH3 expression

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahalingam D, Owonikoko TK, Delpassand E, Mulcahy MF, Kalyan A, Ulahannan S, Cheung K, Izumi Y, Johansen M, Madden T, Shimoyama S, Subach RA, Suzuki T, Wages DS, Wheeler C, Richardson DL. A trial of radiolabeled antibody yttrium-90-FF-21101 for the treatment of advanced ovarian and other cancers. Cancer. 2025 Jan 1;131(1):e35680. doi: 10.1002/cncr.35680. PMID 39748726